CLINICAL TRIAL: NCT02947841
Title: The Effectiveness of Alternating Ventral Intermediate Nucleus Deep Brain Stimulation Parameters in Preventing Tolerance in Essential Tremor Patients
Brief Title: The Effectiveness of Alternating Stimulation in Preventing Tolerance in Essential Tremor Patients
Acronym: AltStim DBS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Oregon Health and Science University (Other)
Responsible Party: Principal Investigator, Shannon Anderson, Movement Disorders Physician Assistant, Oregon Health and Science University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 00015871
Record Dates: First submitted 2016-10-24; First posted 2016-10-28 (Estimated); Last update posted 2018-09-21 (Actual); Status verified 2018-09

CONDITIONS: Essential Tremor; Deep Brain Stimulation
MeSH Terms: conditions — Essential Tremor | interventions — Transcranial Direct Current Stimulation

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Placebo (Placebo Comparator): In the placebo cohort, subjects will alternate their DBS parameters between group A and group B every week for 12 weeks, but they will be blinded to the fact that their group A and group B are equivalent.
  Interventions: Other: Placebo
- Treatment (Active Comparator): In the treatment cohort, subjects will alternate their DBS parameters between group A and group B every week for 12 weeks.
  Interventions: Other: Alternating stimulation

INTERVENTIONS:
Other: Alternating stimulation — Two different, but equally efficacious, settings will be determined for each subject. The settings will differ by a minimum of two of the following parameters: electrode configuration, voltage, frequency and pulse width. The different settings will be named Setting A and Setting B. The treatment cohort will receive both Setting A and Setting B that will differ by the parameters listed above.
  Arms: Treatment
Other: Placebo — The control cohort will receive Setting A but Setting B will be identical to Setting A.
  Arms: Placebo

SUMMARY:
The purpose of this study is to investigate the hypothesis that alternating DBS parameters on a weekly basis will prevent tolerance to stimulation and thus waning of benefit, compared with non-alternating stimulation. The primary endpoint will be preserved tremor control with the alternating group compared with standard treatment using the Tremor Research Group Essential Tremor Rating Assessment Scale (TETRAS). Key secondary endpoints will be preserved activities of daily living measures as well as preserved tremor control as quantified by motion sensor data.

This study has one primary aim: To determine if alternating DBS stimulation parameters on a weekly basis will be superior at preserving tremor control compared with usual stimulation (non-alternating stimulation) in ET patients with VIM DBS.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with clinically diagnosed ET who have had placement of VIM DBS and are willing to undergo a baseline programming visit and 12-week follow-up assessment
2. At least initial benefit from VIM DBS as judged by patient report and clinician exam
3. VIM DBS placement no less than three months from entry into study
4. Patients must demonstrate ability to use patient programmer to switch between group settings on a weekly basis
5. Ability to wear wrist monitor for 2 week intervals, twice during the study 6. Patients with the following IPG types: Activa PC, SC or RC

Exclusion Criteria:

1. Atypical tremor disorder including but not limited to tremor due to multiple sclerosis, medication-induced tremor, Parkinson's disease or parkinsonian syndrome
2. DBS placement complicated by infection, hemorrhage or stroke
3. Previous thalamotomy (either stereotactic, gamma knife or focused ultrasound) or previous DBS surgery resulting in explantation and reimplantation
4. Known incorrect or poor lead placement
5. Inability to change group settings on a weekly basis at least 75% of the time
6. Inability to tolerate 12-week period without additional programming changes, including voltage stimulation adjustment
7. Inability to tolerate 12-week period without adjustment of anti-tremor medications, including primidone, beta-blockers, gabapentin, topiramate and/or benzodiazepines
8. Battery voltage < or equal to 2.70V
9. Patient with the following IPG types: Soletra, Kinetra or Itrel
10. Inability to tolerate two group settings due to side effects or lack of efficacy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 22 (Actual)
Dates: Start 2016-10; Primary Completion 2017-06 (Actual); Study Completion 2017-07 (Actual)

PRIMARY OUTCOMES:
Change from baseline Tremor Research Group Essential Tremor Rating Assessment Scale (TETRAS) performance sub scale at 12 weeks | Through study completion, 12 weeks

SECONDARY OUTCOMES:
Change in TETRAS ADLs scale at 12 weeks | Through study completion, at 12 weeks
Motion sensor data to detect tremor | Two weeks after initial visit; and again at weeks 10-12
  Patients will wear motion sensor device to detect tremor characteristics

CONTACTS AND LOCATIONS:
Overall Officials: Shannon D Anderson, MPAS, PA-C, Principal Investigator — Oregon Health and Science University
Locations (1):
- Oregon Health Science and University, Portland, Oregon, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Baizabal-Carvallo JF, Kagnoff MN, Jimenez-Shahed J, Fekete R, Jankovic J. The safety and efficacy of thalamic deep brain stimulation in essential tremor: 10 years and beyond. J Neurol Neurosurg Psychiatry. 2014 May;85(5):567-72. doi: 10.1136/jnnp-2013-304943. Epub 2013 Oct 4. PMID 24096713
- [Background] Barbe MT, Liebhart L, Runge M, Pauls KA, Wojtecki L, Schnitzler A, Allert N, Fink GR, Sturm V, Maarouf M, Timmermann L. Deep brain stimulation in the nucleus ventralis intermedius in patients with essential tremor: habituation of tremor suppression. J Neurol. 2011 Mar;258(3):434-9. doi: 10.1007/s00415-010-5773-3. Epub 2010 Oct 8. PMID 20927533
- [Background] Zhang K, Bhatia S, Oh MY, Cohen D, Angle C, Whiting D. Long-term results of thalamic deep brain stimulation for essential tremor. J Neurosurg. 2010 Jun;112(6):1271-6. doi: 10.3171/2009.10.JNS09371. PMID 19911883
- [Background] Shih LC, LaFaver K, Lim C, Papavassiliou E, Tarsy D. Loss of benefit in VIM thalamic deep brain stimulation (DBS) for essential tremor (ET): how prevalent is it? Parkinsonism Relat Disord. 2013 Jul;19(7):676-9. doi: 10.1016/j.parkreldis.2013.03.006. Epub 2013 Apr 11. PMID 23582712
- [Background] Pilitsis JG, Metman LV, Toleikis JR, Hughes LE, Sani SB, Bakay RA. Factors involved in long-term efficacy of deep brain stimulation of the thalamus for essential tremor. J Neurosurg. 2008 Oct;109(4):640-6. doi: 10.3171/JNS/2008/109/10/0640. PMID 18826350